CLINICAL TRIAL: NCT02170389
Title: Neoadjuvant AGS-003 Immunotherapy in Patients With Localized Kidney Cancer <pT2
Brief Title: Vaccine Therapy Before Surgery in Treating Patients With Localized Kidney Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor having financial difficulties
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 250113; NCI-2014-01254 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AGS-003-012; I 250113 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Recurrent Renal Cell Carcinoma; Stage I Renal Cell Cancer; Stage II Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nephrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (AGS-003 immunotherapy, nephrectomy) (Experimental): Patients receive 3 injections of renal cell carcinoma/cluster of CD40L RNA-transfected autologous dendritic cell vaccine AGS-003 ID once every 7 days during weeks 6-8 in the absence of disease progression or unacceptable toxicity. Patients then undergo partial or radical nephrectomy on week 10.
  Interventions: Other: Laboratory Biomarker Analysis; Procedure: Nephrectomy; Biological: Renal Cell Carcinoma/CD40L RNA-Transfected Autologous Dendritic Cell Vaccine AGS-003

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Nephrectomy — Undergo partial or radical nephrectomy
Biological: Renal Cell Carcinoma/CD40L RNA-Transfected Autologous Dendritic Cell Vaccine AGS-003 — Given ID
  Other Names: AGS-003

SUMMARY:
This pilot clinical trial studies vaccine therapy before surgery in treating patients with kidney cancer that has not spread to nearby lymph nodes or to other parts of the body. Vaccines made from a person's tumor cells and white blood cells may help the body build an effective immune response to kill tumor cells when they are infused back into the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the immune-modulatory systemic and intratumoral effects of AGS-003 (renal cell carcinoma/cluster of differentiation [CD]40L ribonucleic acid [RNA]-transfected autologous dendritic cell vaccine AGS-003) as neoadjuvant treatment in patients with localized renal cell carcinoma.

SECONDARY OBJECTIVES:

I. To assess the feasibility that total tumor RNA processing-related activities meet specifications for AGS-003 manufacturing utilizing a core needle biopsy procedure for tumor harvesting prior to nephrectomy.

OUTLINE:

Patients receive 3 injections of renal cell carcinoma/cluster of CD40L RNA-transfected autologous dendritic cell vaccine AGS-003 intradermally (ID) once every 7 days during weeks 6-8 in the absence of disease progression or unacceptable toxicity. Patients then undergo partial or radical nephrectomy on week 10.

After completion of study treatment, patients are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Have localized non-metastatic renal cell carcinoma (RCC) (< pT2, NO, MO), as per the American Joint Committee on Cancer (AJCC) seventh (7th) edition criteria
* Must be surgical candidates as deemed fit by surgeon
* Patients of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform the treating physician immediately
* Willingness to undergo leukapheresis and biopsy procedures for the autologous components (peripheral blood mononuclear cells, plasma and fresh tumor specimen) required for manufacture of AGS-003
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (e.g., shortness of breath, fatigue, orthopnea, paroxysmal nocturnal dyspnea), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Radiation to primary tumor prior to enrollment in this study
* Pregnant or nursing female patients
* Unwilling or unable to follow protocol requirements
* Active autoimmune disease or condition requiring chronic immunosuppressive therapy (e.g., rheumatoid arthritis, systemic lupus erythematous, multiple sclerosis, organ transplant recipient, etc.)

  * NOTE: abnormal laboratory values for autoimmunity markers in the absence of other signs/symptoms of autoimmune disease are not exclusionary
* Known clinically significant infections, including human immunodeficiency virus (HIV) and active hepatitis B or C
* Any condition which in the Investigator's opinion deems the patient an unsuitable candidate to receive treatment (i.e., any significant medical illness or abnormal laboratory finding that would, in the investigator's judgment, increase the subject's risk by participating in this study)
* Chronic use of systemic corticosteroids (i.e., >= 10 mg/day prednisone or equivalent)
* Received an investigational agent within 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-10-14 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. med.Thomas Schwaab, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (AGS-003 Immunotherapy, Nephrectomy)
Started | 5
Completed | 4
Not Completed | 1
Not completed — Study terminated prior to start of treat | 1

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Treatment (AGS-003 Immunotherapy, Nephrectomy)
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (19.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Immune Marker Expression [Mean (Standard Deviation); unit: units on a scale] — Population: Pre and post treatment samples were to be analyzed in batch. The study was terminated early due and samples were not analyzed.

OUTCOME MEASURES:

1. Primary Outcome: Change in Immune Marker Expression Levels
Description: The time component will be modeled as a three-level classification factor. The full model for the effects of time will be fit using linear mixed model methods. The model will include a random patient effect and 5 fixed effects for time and the interactions. The presence of any time effect will be assessed with full-reduced model type 3 test. If the omnibus test is statistically significant at the p < 0.05 level, then three pairwise time-point comparisons will be conducted.
  Expression measurements may be transformed to satisfy modeling assumptions.
Time Frame: Baseline to up to 30 days post-nephrectomy
Population: The clinical trial was terminated due to lack of funding before data were collected.
Arm/Group | Treatment (AGS-003 Immunotherapy, Nephrectomy)
Number analyzed (Participants) | 0

2. Secondary Outcome: Adverse Event Rates as Graded by the Common Terminology Criteria for Adverse Events Version 4.0
Description: Summarized in all patients who received AGS-003. These rates will be described as the proportion of patients with the event, by grade, and supported with exact 95% confidence intervals.
Time Frame: Up to 30 days
Population: Only patients who received any injections were included.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Treatment (AGS-003 Immunotherapy, Nephrectomy)
Number analyzed (Participants) | 4
percentage of subjects
  Any Grade AE | 100 [40 to 100]
  Any Grade 1 | 100 [40 to 100]
  Any Grade 2 | 50 [7 to 93]
  Any Grade 3 | 25 [5 to 70]
  Any Grade 4 | 0 [0 to 49]
  Any Grade 5 | 0 [0 to 49]

ADVERSE EVENTS:
Time Frame: All deaths and new AEs occurring from the date of signed consent until 30-days after the administration of the last study treatment or a new treatment is started, are reported.
Arm/Group | Treatment (AGS-003 Immunotherapy, Nephrectomy)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (AGS-003 Immunotherapy, Nephrectomy) (N=4)
Bundle branch block (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Inflammation (General disorders) | 1 (2)
Influenza like illness (General disorders) | 1 (1)
Injection site inflammation (General disorders) | 1 (1)
Injection site pain (General disorders) | 1 (1)
Injection site pruritus (General disorders) | 1 (1)
Injection site reaction (General disorders) | 2 (2)
Injection site swelling (General disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (2)
Procedural pain (Injury, poisoning and procedural complications) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT02170389/Prot_SAP_001.pdf